CLINICAL TRIAL: NCT03341624
Title: Surgical Treatment and Prognosis of Congenital Cataract With Persistent Fetal Vasculature
Brief Title: Congenital Cataract With Persistent Fetal Vasculature
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HM-PFV-001
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Persistent Fetal Vasculature; Congenital Cataract
Keywords: persistent fetal vasculature; congenital cataract
MeSH Terms: conditions — Persistent Hyperplastic Primary Vitreous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cataract surgery cataract extraction and intraocular implanta (Experimental)
  Interventions: Procedure: cataract surgery cataract extraction and intraocular implantation

INTERVENTIONS:
Procedure: cataract surgery cataract extraction and intraocular implantation

SUMMARY:
To observe the clinical characteristics and surgical treatment of 24 cases of congenital cataract complicated with Persistent Fetal Vasculature (PFV) in 28 cases of congenital cataract in our hospital.

DETAILED DESCRIPTION:
methods the clinical data of 28 eyes of 24 children with congenital cataract complicated with PFV who underwent surgical treatment in our hospital were analyzed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* congenital cataract with Persistent Fetal Vasculature

Exclusion Criteria:

* congenital cataract with no Persistent Fetal Vasculature

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 2 years
  level1：visual acuity≥0.3；level 2：0.1≤visual acuity<0.3；level 3：0.02 ≤visual acuity<0.1；level 4：≤0.02

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No